CLINICAL TRIAL: NCT02130297
Title: Post Excision/Mohs Fractional CO2 Resurfacing: A Quantitative and Qualitative Scar Analysis Study
Brief Title: Post Excision/Mohs Scar Laser Resurfacing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Hooman Khorasani, Clinical Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GCO 14-0387
Record Dates: First submitted 2014-04-29; First posted 2014-05-05 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Skin Cancer
Keywords: Mohs; scar; post excision; CO2 laser; laser; skin cancer; resurfacing
MeSH Terms: conditions — Skin Neoplasms; Cicatrix | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 - day 1 (Active Comparator): Group 1 will receive laser therapy to half of the scar the day of the excision.
  Interventions: Device: Laser Treatment
- Group 2 - day 14 (Active Comparator): Group 2 will receive laser therapy at the time of suture removal or post-operative day 14.
  Interventions: Device: Laser Treatment
- Group 3 - week 9 (Active Comparator): Group 3 will receive laser treatment to half the scar at the 9 week postop visit.
  Interventions: Device: Laser Treatment

INTERVENTIONS:
Device: Laser Treatment — The subject will receive ablative fractional resurfacing with the Deep and Active FXTM platforms of the Lumenis Ultrapulse CO2 laser. The settings for treatment of scars on the face with the Deep platform will be 15% coverage, 15mJ at 150 Hz and 15% coverage, 12.5 mJ at 150 Hz for off the face. The Active platform settings will be 90 mJ with a density of 3 for the face and 70 mJ and a density of 2 for off the face. The DeepFXTM platform will be applied to the scar prior to the ActiveFX TM platform. Half of the excision scar will be treated with the appropriate settings and half will go untreated.
  Other Names: Lumenis UltraPulse Total FXTM fractionated CO2 laser

SUMMARY:
The purpose of this study is to evaluate the potential benefits of treating a surgical scar post excision with an ablative fractionated CO2 laser with the goal of decreasing the appearance and size of the scar.

DETAILED DESCRIPTION:
The objective of this research is to determine, through a split scar study, that treating a post excision scar with a fractionated ablative CO2 laser improves both the texture and cosmetic appearance of the scar. An attempt will be made to determine the ideal timing for treating the excision scar as previous studies have ranged from treating the day of the excision up till 10 weeks post-excision. In order to evaluate the treated portion versus untreated portion of the scar, investigators and the subjects will use a quartile rating scale. In addition, punch biopsy samples will be taken to quantify the difference in collagen architecture 9 weeks after treatment with the laser.

There will be a total of 7 study visits to include the day of the excision and laser treatment if randomized to this group, post-op day number 14 for suture removal as well as laser therapy if the subject has been randomized to that treatment group, 4 weeks post-op, 9 weeks post-op and laser treatment for subjects randomized to this time frame for treatment, 12 weeks post-op, 17 weeks post-op and 24 weeks post-op. Each visit will last approximately 30-45 minutes each in which clinical photos of the surgical scar will be taken and any wound care or side effects of the laser therapy or surgery will be addressed. Healing and scar appearance will be reviewed and rated at each of the six postsurgical visits.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form.
* Must be male or female and aged >18 years at the time of consent.
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Patients undergoing skin excisions of the face/trunk/extremities.

Exclusion Criteria:

* Inability to provide voluntary informed consent
* Use of laser or light based treatments to affected areas in past year
* Fitzpatrick Skin types 3-5
* Surgical lesions located on the central chest
* History of keloid formation
* History of Accutane in the last six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hooman Khorasani, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Original protocol had 3 arms. Due to difficulty with enrollment, study did not perform a laser treatment at 9 weeks and the enrolled participants were all given the same intervention.
Groups:
- Participants With Fitzpatrick Skin Phototype I or II: Participants with wounds to limbs of Fitzpatrick skin phototype I or II to receive laser therapy to half of the scar the day of the excision, Day 0; and to the other half on Day 14.
Period: Overall Study
Arm/Group | Participants With Fitzpatrick Skin Phototype I or II
Started | 30
Completed | 26
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Fitzpatrick Skin Phototype I or II
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 56 [34 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Scar length [Mean (Full Range); unit: cm] | 6.4 [3.6 to 12.6]

OUTCOME MEASURES:

1. Primary Outcome: MMSS for Scar Halves Treated
Description: modified Manchester scar scale (MMSS) treated - Full scale from 5 to 18, with higher score indicating lower health outcomes
Time Frame: Day 0 and Day 14
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Participants With Fitzpatrick Skin Phototype I or II
Number analyzed (Participants) | 26
score on a scale
  Day 0 | 8.4 [7 to 10]
  Day 14 | 8.7 [7 to 11]

2. Secondary Outcome: Quantitative Scar Analysis as Measured by Fractal Dimension (Fd) and Lacunarity
Description: Fd indicates scar tissue density - a measure of how completely an object fills space and increases in value with increasing structural density. It has a value between 1 and 2: a minimum value of 1 corresponds to a straight line filling the space, and a maximum value of 2 corresponds to an object completely occupying the entire space.
  Lacunarity describes the characteristics of fractals of the same dimension with different texture appearances and indicates scar tissue architecture (homogeneous vs. heterogeneous) - a measure of the nonuniformity (heterogeneity) of a structure or the degree of structural variance within an object. L has a value between 0 and 1, where a minimum value of 0 corresponds to an absolute homogeneous object.
Time Frame: Day 0 and Day 14
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Participants With Fitzpatrick Skin Phototype I or II
Number analyzed (Participants) | 30
units on a scale
  Fractal dimension (Fd) Day 0 | 1.778 [1.691 to 1.830]
  Fractal dimension (Fd) Day 14 | 1.781 [1.706 to 1.831]
  Lacunarity Day 0 | 0.368 [0.225 to 0.637]
  Lacunarity Day 14 | 0.345 [0.214 to 0.573]

3. Secondary Outcome: Quartile Scale
Description: Comparison of scars using quartile scale: 0 indicates no difference, 1 indicates a 1-25% difference or "mild" difference, 2 indicates a 26-50% or moderate difference, 3 indicates a 51-75% or significant improvement and 4 indicates a 76-100% difference or very significant.
Time Frame: 24 weeks post-op
Population: Data not collected
Arm/Group | Participants With Fitzpatrick Skin Phototype I or II
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Participants With Fitzpatrick Skin Phototype I or II
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 20/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Fitzpatrick Skin Phototype I or II (N=26)
transient erythema (Skin and subcutaneous tissue disorders) | 20
swelling and crusting (Skin and subcutaneous tissue disorders) | 20

LIMITATIONS AND CAVEATS:
Single-center study with wounds limited to limbs of skin phototype I-II subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT02130297/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT02130297/SAP_001.pdf